CLINICAL TRIAL: NCT02204852
Title: Safety and Efficacy of Iloprost and Eptifibatide Co-administration Compared to Standard Therapy in Patients With Septic Shock - a Randomized, Controlled, Double-blind Investigator-initiated Trial
Brief Title: Co-administration of Iloprost and Eptifibatide in Septic Shock Patients
Acronym: CO-ILEPSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sisse R. Ostrowski, MD PhD DMSc (Other)
Responsible Party: Sponsor-Investigator, Sisse R. Ostrowski, MD PhD DMSc, MD, PhD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO-ILEPSS
Record Dates: First submitted 2014-07-24; First posted 2014-07-30 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iloprost+eptifibatide (Experimental): Co-administration of 1 ng/kg/min Ilomedin® and 0.5 µg/kg/min Integrilin® as 48h continuous i.v infusions
  Interventions: Drug: Iloprost+eptifibatide
- Saline (Placebo Comparator): Double dummy 0.9% saline as 48h continuous i.v infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iloprost+eptifibatide
  Other Names: Ilomedin(R); Integrilin(R)
  Arms: Iloprost+eptifibatide
Drug: Placebo
  Other Names: 0.9% saline, double dummy
  Arms: Saline

SUMMARY:
Objective Evaluating the safety and efficacy of iloprost and eptifibatide co-administration compared to placebo as an addition to standard care in septic shock patients.

Trial rationale Iloprost and eptifibatide combination therapy in septic shock patients is expected to deactivate the endothelium and restore vascular integrity, reduce formation of microvascular thrombosis and dissolve existing clots in the microcirculation and maintain platelet counts, thereby improving platelet-mediated immune function and reducing the risk of bleeding. Together this is expected to translate into reduced organ failure and improved outcome in patients with septic shock.

Trial population The trial population is patients >18 years admitted to the ICU with septic shock within the last 24h. Eighteen evaluable septic shock patients will be included.

Trial design This is a single center, randomized (2:1, active:placebo), placebo controlled, double-blind investigator-initiated phase IIa trial in patients with septic shock, investigating the safety and efficacy of co-administration of Iloprost and Eptifibatide as a 48h continuous i.v infusion in totally 18 patients.

All patients will receive standard ICU care including LMWH thrombosis prophylaxis.

As all patients present at the trial site in an acute, critical condition, scientific guardians will co-sign the informed consent form before inclusion. Next-of-kin and the patients' general practitioner will co-sign as soon as possible and the patient will provide informed consent whenever possible. The active treatment is expected to improve the clinical condition of the individual patient and to provide information that may translate into improved therapy of future sepsis patients.

During the study, blood samples will be taken at different time points. Patients will be observed and assessed continuously with regards to complications including bleeding. Patients will be actively assessed as long as the patient is in the ICU. During the extended follow up period at day 30 and 90, contact will be made with the patients to follow up on safety events and vital status.

The trial is conducted in accordance with the protocol and the current regulatory requirements and legislation in Denmark.

Investigational product The active treatment in the trial comprises co-administration of 1 ng/kg/min Ilomedin® and 0.5 µg/kg/min Integrilin® as 48h continuous i.v infusions. The drugs will be purchased and administered according to the product specifications.

Placebo The placebo in the trial is 0.9% saline as 48h continuous i.v infusion, which will be used as placebo for both study drugs. The i.v volume of placebo saline to be administered is equal to the administered volume of diluted (in 0.9% saline) active drug.

Data protection In compliance with the Danish data protection law, the trial will be approved by the Danish Data Protection Agency.

Sponsor of study and financial support This research project is investigator-initiated by the trial sponsor and co-investigator Sisse R. Ostrowski and co-investigator Pär I. Johansson in collaboration with the principal investigator Morten Bestle.

It has not received funding from any commercial sponsors.

Time line Patient recruitment period runs from September 2014 to August 2015. Follow-up data on 30-day and 90-day outcome and adverse events will be collected. Initial data analyses will be done after completion of 30-day follow-up for all patients. Secondary data analyses will be done after completion of 90-day follow-up for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult intensive care patients (age ≥18 years) AND
2. Sepsis, defined as suspected or confirmed site of infection or positive blood culture and ≥2 of 4 systemic inflammatory response syndrome (SIRS) criteria fulfilled within the last 24h:

   * Temperature ≤ 36˚ C or ≥ 38˚C
   * Heart rate ≥ 90 beats per minute
   * Mechanical ventilation for acute respiratory process or respiratory rate ≥ 20 breaths per minute or PaCO2 < 4.2 kPa
   * WBC ≥ 12,000/mm³ OR ≤ 4,000/mm³ OR > 10% bands AND
3. Septic shock within the last 24h, defined as:

   * Hypotension (MAP <70 mmHg, Lactate 4 mmol/L) despite ongoing resuscitation with fluids (crystalloids, colloids, blood products) within the last 24h OR
   * ≥30 ml/kg ideal body weight (IBW) fluid (crystalloids, colloids, blood products) given in the last 24h AND
   * Need for vasopressor/inotropic agents (noradrenaline, adrenaline, dopamine) within the last 24h AND
4. Can be randomized into trial and dosed < 24h after septic shock diagnosis (the time-point for the septic shock diagnosis corresponds to the time-point where the vasopressor/inotropic therapy (3c) is initiated) AND
5. Consent is obtainable

Exclusion Criteria:

1. Patient is pregnant or breast-feeding
2. Patient weights more than 125 kg
3. Patients with known allergy towards any of the investigational products or contraindications which should be excluded according to the investigational product specifications
4. Patients in whom the clinician finds antithrombotic therapy contraindicated - prophylaxis included
5. Patients at increased risk of bleeding:

   * Surgery in the previous 48h and expected surgery within 48 h
   * Epidural or spinal puncture in the previous 12h
   * Platelet count less than 10,000/mm3 in the previous 24h
   * Need of blood products for bleeding in the previous 24h (3 or more RBC/24 h)
   * Treatment with any antithrombotics within 12h (profylaxis excepted)
   * Current intracranial bleeding
   * Traumatic brain or spinal injury within the last month
6. Patients requiring any form of antithrombotics (beyond profylaxis) in therapeutic doses or prothrombotics in any dose, including:

   * Unfractionated heparin within 8h before the infusion (prophylactic heparin up to 15,000 U/day permitted)
   * LMWH within 12h before the infusion (prophylactic doses permitted)
   * Warfarin within 1 day before the infusion
   * Acetylsalicylic acid more than 650 mg/day within 3 days before the study
   * Thrombolytic therapy within 3 days before the study (catheter clearance doses permitted)
   * GPIIb/IIIa receptor inhibitors within 4 days before the study
   * Antithrombin III with dose greater than 10,000 U within 12h before the study
7. Patients with a do-not-resuscitate order (expected not to survive more than few days because of uncorrectable medical or surgical condition other than sepsis)
8. Patient with chronic renal failure requiring dialysis (renal failure without need for dialysis permitted)
9. Patients who have undergone transplantation of bone marrow, liver, pancreas, heart, lung, or bowel (kidney transplant permitted)
10. Patient with known hypercoagulable condition:

    * Activated protein C resistance
    * Hereditary protein C, protein S, or antithrombin III deficiency
    * Anticardiolipin or antiphospholipid antibody
    * Lupus anticoagulant
    * Homocysteinemia
    * Recent or highly suspected pulmonary embolism or deep venous thrombosis (within 3 months)
11. Patients with known congenital hypocoagulable diseases
12. Patient with known primary pulmonary hypertension

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Mean change i plasma biomarkers reflecting endothelial damage | 48 hours
  Change in biomarkers indicative of endothelial activation and damage (sE-selectin, syndecan-1, thrombomodulin, sVE-cadherin, nucleosomes) from baseline to 48 hours post-randomization
Mean change in platelet count reflecting platelet consumption | 48 hours
  Change in platelet count from baseline to 48 hours post-randomization
Mean change in biomarkers reflecting fibrinolysis | 48 hours
  Change in D-dimer and fibrin split products indicative of fibrinolysis (fibrinogen degradation Bβ15-42; fibrin degradation Fragments X, Y, D and E) from baseline to 48 hours post-randomization

SECONDARY OUTCOMES:
Number of patients with severe bleeding | 24 hours to 90 days
  Severe bleeding (intracranial or clinical bleeding with the use of 3 RBC units or more/24 hours)
Number of patients with transfusion requirements | 24 hours to 90 days
  Use of blood products (in ICU) post-randomization
Mortality | 7 to 90 days
  Difference in day 7, 30 and 90 day mortality between patients receiving active treatment (eptifibatide and iloprost) and placebo
Mean change in disease severity score | 48 hours to 7 days
  Changes in SOFA score from baseline to 48 h and day 5 and 7 post-randomization
Number of patients requiring organ support | 48 hours to 90 days
  Days of vasopressor, ventilator and renal replacement therapy post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Sisse R Ostrowski, MD, PhD, DMSc, Study Chair — Copenhagen University Hospital, Rigshospitalet, Denmark; Pär I Johansson, MD, DMSc, MPA, Study Director — Copenhagen University Hospital, Rigshospitalet, Denmark
Locations (1):
- Department of Anesthesia and Intensive Care, Nordsjællands Hospital, Hillerød, Capital Region, Denmark

REFERENCES:
- [Derived] Berthelsen RE, Ostrowski SR, Bestle MH, Johansson PI. Co-administration of iloprost and eptifibatide in septic shock (CO-ILEPSS)-a randomised, controlled, double-blind investigator-initiated trial investigating safety and efficacy. Crit Care. 2019 Sep 5;23(1):301. doi: 10.1186/s13054-019-2573-8. PMID 31488213